CLINICAL TRIAL: NCT02558985
Title: Pulmonary Compliance Changes During Manipulation of Early Onset Scoliosis and Cast
Brief Title: Pulmonary Compliance Changes During Manipulation of Early Onset Scoliosis and Cast Application
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Tyler William Christman, Orthopaedic Surgeon, Indiana University
Other Study IDs: 1503944048
Record Dates: First submitted 2015-08-29; First posted 2015-09-24 (Estimated); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Scoliosis
Keywords: Pulmonary Compliance; Casting
MeSH Terms: conditions — Scoliosis; Patient Compliance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Casting — Serial casting is used to partially correct the deformity before beginning bracing. A cast can be considered a full-time brace which cannot be removed.

SUMMARY:
No interventions outside the normal course of patient care. The investigators will be collecting data at specified points throughout the casting process.

The proposed study will measure lung compliance during the casting process for spinal manipulation. Research questions include: Is there a quantifiable change in lung compliance during the casting process? Is there an individual change in lung compliance over time comparing collection points at each cast change? Is there a change in appearance of flow-volume loop? Is there a decrease in oxygen saturation from post-induction baseline? The investigators hypothesize that there is a change in lung compliance and a decrease in oxygen saturation during the casting process.

DETAILED DESCRIPTION:
All patients undergoing spine manipulation and scoliosis casting will receive general anesthesia with a standard anesthetic technique regardless of if the patient is included in the study or not. The investigators will meet with the patient and the patient's parent/guardian prior to the procedure, which is traditionally done whether a patient participates in a study or not, to discuss the anesthetic plan. As part of the investigator's description of the anesthetic plan, the investigator will inform the patient and the parent/guardian of the study including the rationale for the study and the non-invasive means of obtaining data. The data will be obtained during the current cast application as well as any subsequent cast application surgeries that the patient will return for the future. A patient's cast will be changed approximately as needed per each child's circumstance; common time periods a child's cast may need to be changed include, but not limited to: growth, the cast becoming soiled, damaged, or other circumstances the study physician feels it is advisable to change the cast. The study will follow them until casting procedures are completed for treatment of scoliosis. The standard general anesthesia technique will be used. Please see Appendix A for suggested Anesthesia.

There will be seven data collection points during the patient's general anesthetic:

1. Prior to the removal of the old cast, if applicable
2. After removal of old cast, if applicable
3. In frame, pre-traction
4. In frame, in traction
5. Post-body cast application (prior to cast windows; in traction)
6. Post cast application in bed out of traction (prior to cutting out windows)
7. Post-cast windows cut out (in bed, prior to return of spontaneous ventilation)

The data collection will include the following physiologic parameters:

1. Non-invasive blood pressure
2. Heart rate
3. Oxygen saturation
4. The amount of traction (in pounds) that the patient is placed in for the spine manipulation. This will be measured at the beginning of traction, the beginning of cast application, and at the end of cast application.
5. Respiratory measurements from the Philips Spirometry Module, consisting of:

   1. lung compliance
   2. tidal volume
   3. peak inspiratory pressure
   4. flow volume loop
   5. airway resistance

Patients will also be subject to a chart review. The chart review will include previous anesthetic records which may provide valuable information concerning the patient's baseline lung compliance, tidal volume, peak inspiratory pressure, flow volume loop, and airway resistance, amount of traction applied and scoliosis curve correction. This previous data will be used to compare to the data collected before, during and after cast changes.

Appendix A: Suggested Anesthesia

1. Premedication: 0.5mg/kg midazolam PO (max 15mg), PRN
2. Induction: Mask with sevoflurane in oxygen
3. Secure Intravenous Access
4. Intubation: Propofol 3-4mg/kg IV. Oral endotracheal tube.
5. Ventilation: Controlled using volume mode at 8ml/kg
6. Maintenance: oxygen, sevoflurane, controlled ventilation
7. Emergence: ondansetron 0.15mg/kg IV

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Progressive Early Onset Scoliosis
* 6 months to 9 years of age
* Must be able to present for serial thoracolumbar casting and spine manipulation at Riley Hospital for Children in Indianapolis, IN

Exclusion Criteria:

• Known contraindication to the general anesthesia

Ages: 6 Months to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Any patients 6 months to 9 years of age with progressive Early Onset Scoliosis who present for serial thoracolumbar casting and spine manipulation at Riley Hospital for Children will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Change in lung parameters for an individual patient as his/her own control During each casting and the duration of casting treatment. | up to 60 months
  Change in lung parameters for an individual patient as his/her own control, during the casting application as well as serial compliance measurements during the course of the casting treatment in both the acute and long-term phase of casting and the duration of casting. Parameters measured would include, but not limited to lung compliance, tidal volume, peak inspiratory pressure, flow volume loop, and airway resistance.

SECONDARY OUTCOMES:
Measure the oxygen saturation from post-induction baseline during the casting application as well as serial compliance measurements | up to 60 months
  Measure the percent of oxygen saturation to determine if there is a difference between initial cast application and subsequent cast applications.

OTHER OUTCOMES:
Change in appearance of flow-volume loop | up to 60 months
  Change in appearance of flow-volume loop, during the casting application as well as serial compliance measurements during the course of the casting treatment
  Change in appearance of flow-volume loop, during the casting application as well as serial compliance measurements during the course of the casting treatment
Correlate the change in compliance with the amount of traction applied during the casting application | up to 60 months
  (in respiratory physiology) a measure of distensibility of the lung volume produced by a unit pressure change with the amount of pounds of traction applied.
Compare scoliosis casting patient data to healthy patients' lung compliance, during the casting application as well as serial compliance measurements during the course of the casting treatment | up to 60 months
  Comparison of Respiratory measurements from the Philips Spirometry Module, consisting of: lung compliance, tidal volume, peak inspiratory pressure, flow volume loop, airway resistance in Scoliosis Patients compared to healthy normal patients

CONTACTS AND LOCATIONS:
Overall Officials: Tyler W Christman, DO, Principal Investigator — Indiana University
Locations (1):
- Riley Hospital, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Mehta MH. Growth as a corrective force in the early treatment of progressive infantile scoliosis. J Bone Joint Surg Br. 2005 Sep;87(9):1237-47. doi: 10.1302/0301-620X.87B9.16124. PMID 16129750
- [Background] Jensen RD: Cardiorespiratory Effects of Derotational Casting during Anesthesia for Children with Early Onset Scoliosis4: 36-40, OJA, 2014